CLINICAL TRIAL: NCT02729922
Title: Registry of Patients With CardioMEMS
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 824716
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cardiomems — Eligible patients will undergo implantation of a pulmonary artery sensor (CardioMEMS), a wireless implantable hemodynamic monitoring system in the cardiac catheterization laboratory. This system has a passive wireless, radiofrequency sensor without batteries or leads. Patients transmit data through a device in their home that interacts wirelessly with the sensor. Clinicians retrieve this data via a web interface to use in making management decisions for patients.

SUMMARY:
CardioMEMS is an implantable wireless hemodynamic monitoring system which can transmit the pulmonary artery pressure. This device is FDA approved to be used as a diagnostic tool to help management of selected heart failure patients. Heart failure patients with NYHA class III heart failure, irrespective of the left ventricular ejection fraction, and a previous hospital admission for heart failure in the past 12 months, without stage IV or V chronic kidney disease are candidates to receive a CardioMEMS device. Our goal is to create a registry of all patients that receive a CardioMEMS device and monitor outcomes, primarily heart failure hospitalizations, heart failure related quality of life and re-admissions.

DETAILED DESCRIPTION:
Background Clinical trials with CardioMEMS were done and the device is now FDA approved for use in heart failure patients with NYHA class III heart failure for at least three months, irrespective of the left ventricular ejection fraction, with a previous hospitalization for heart failure in the last 12 months. Patients with chronic kidney disease stage IV or V are excluded.

Briefly, the CHAMPION Trial, which was published in the Lancet (Lancet 2011; 377: 658-66), enrolled patients in 64 centers in the USA and were randomly assigned by the use of a centralized electronic system to management with CardioMEMS or a control group. The patients were followed for six months. The treatment group used daily measures of pulmonary artery pressures in addition to standard of care versus standard of care alone in the control group. The protocol for the treatment group was to lower the pulmonary artery pressures when elevated, using neurohormonal, diuretic, or vasodilator drugs. The control group continued to have drug changes in response to patients' clinical signs and symptoms rather than the pulmonary artery pressure. All patients were on optimum drug and device therapies at the time of sensor implantation in accordance to the ACC and AHA guidelines. At six months the treatment group had a 37% reduction in heart failure related hospitalizations, patients with more days alive outside the hospital, and better quality of life compared to the control group.

A follow up study was published in the Lancet (Lancet 2016; 387:453-461) which examined the extended efficacy of this strategy over 18 months looking at the clinical effect of open access to pressure information and monitored the original treatment group for an additional 13 months. After pulmonary artery pressure information became available to guide therapy during open access (the devices in the control group were activated and followed for the 13 months after the initial six months), rates of admissions to hospital for heart failure in the former control group were reduced by 48% compared with rates of admissions in the control group during randomized access (initial six months).

These studies show that both short term and long term management of NYHA Class III heart failure based on home transmission of pulmonary artery pressure with an implanted pressure sensor has significant short-term and long-term benefit in lowering hospital admission rates for heart failure.

Patients aged 18 years or older with moderate NYHA functional class III heart failure for at least 3 months, irrespective of left ventricular ejection fraction or cause, and a hospitalization for heart failure within the past 12 months are eligible for a CardioMEMS device. If the patient is thought to be a good clinical candidate, with difficult to manage fluid status, the patient and their Heart Failure Cardiologist will discuss the option of having a CardioMEMS device implanted for standard of care treatment. If the device is implanted, the patient will be asked to be enrolled in the registry. The patient will have normal clinical follow up and clinically standard interrogations. The device interrogations will be sent daily from the patient and reviewed once a week unless the patient calls with symptoms or weight gain in which it will be reviewed at that time. If changes in medications are made, the patient's device will be interrogated daily for 3 subsequent days and then return to the baseline weekly interrogation. The data obtained from the interrogation is the pulmonary artery pressure. There are no research interventions outside of normal standard clinical care. All of the clinically collected data will be recorded in the Penn CardioMEMS registry.

Patients will be followed up in clinic one month after implant, then 3 months and then as determined by their Heart Failure Cardiologist as part of usual clinical care. A quality of life assessment will be done at each clinic appointment for the first year (Minnesota Living with Heart Failure questionnaire).

Adverse events will be recorded as they occur. There are device-related or system-related complications such as bleeding complications or pressure-sensor failures defined as the inability to obtain recordings. Of note, during the clinical trials there were no pressure-sensor failures.

The data will be collected from the clinical electronic medical record and administrative data sets at the University of Pennsylvania.

Standard statistical methods will be used. Statistical analysis will be done with Wilcoxon rank sum test and student's t test with alpha=0.05. Patient survival rates will be analyzed by Kaplan-Meier method and the log-rank test.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* NYHA class III heart failure
* Heart Failure Hospitalization in the last 12 months
* Optimal heart failure medical and device therapies per national heart failure guidelines

Exclusion Criteria:

* History of recurrent pulmonary embolism or deep vein thrombosis
* Cardiac resynchronization device placement in the last three months
* Stage IV or V chronic kidney disease
* Unable to take anti-platelet or anti-coagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with New York Heart Association functional class III heart failure for at least three months, irrespective of left ventricular ejection fraction or cause, and a hospitalization for heart failure within the past 12 months who are on optimal medical and device management. Patients being referred for the placement of a Cardiomems device by their clinical Heart Failure Cardiologist will be invited to participate in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2025-06 (Actual); Study Completion 2025-06 (Actual)

PRIMARY OUTCOMES:
Heart Failure Hospitalizations | 1 year
  Number of admissions to the hospital for the treatment of heart failure

SECONDARY OUTCOMES:
Heart Failure Related Quality of Life | 1 year
  Minnesota Living with Heart Failure Questionaire

OTHER OUTCOMES:
Heart Failure Outpatient Visits | 1 year
  Number of outpatient visits to monitor or treat heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Lee R Goldberg, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abraham WT, Adamson PB, Bourge RC, Aaron MF, Costanzo MR, Stevenson LW, Strickland W, Neelagaru S, Raval N, Krueger S, Weiner S, Shavelle D, Jeffries B, Yadav JS; CHAMPION Trial Study Group. Wireless pulmonary artery haemodynamic monitoring in chronic heart failure: a randomised controlled trial. Lancet. 2011 Feb 19;377(9766):658-66. doi: 10.1016/S0140-6736(11)60101-3. PMID 21315441